CLINICAL TRIAL: NCT06152562
Title: Evaluation of Platelet Therapy Response in Left Ventricular Assist Device Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Thomas Schlöglhofer, VAD Engineer, Medical University of Vienna
Other Study IDs: EK Nr: 2460/2020; 2021-004921-62 (EudraCT Number)
Record Dates: First submitted 2021-12-10; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: End-stage Heart Failure; Cardiomyopathies; Mechanical Circulatory Support
Keywords: Left ventricular assist device
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individualized ASA therapy group using platelet inhibition monitoring: The first VerifyNow ARU measurement will be done minimum 2 hours and at latest 24 hours after the first four doses of ASA. If the ARU is ≤ 549, the current daily ASA dose will be continued and the patient will be discharged with this dose. If the ARU is ≥ 550, the dose will be increased by 50 mg and the test is repeated after two doses. We will increase the dose step by step until the ARU decreased below 550 or a maximum ASA dose of 300 mg per day is reached. If there is no sufficient drug effect at the maximum dose assessed by VerifyNow, the patient will be count as non-responder and a change to a P2Y12-inhibitor (e.g. Clopidogrel 75 mg) is indicated. A resistance against Clopidogrel will not be examined. The other tests will be held at the first follow-up visit and six months after implantation.
  Interventions: Diagnostic Test: VerifyNow antiplatelet therapy response test
- Standard ASA therapy: Initiation of standard dose ASA therapy as per center guidelines with HeartMate 3: 100mg/day; HVAD: 200mg/day

INTERVENTIONS:
Diagnostic Test: VerifyNow antiplatelet therapy response test — VerifyNow testing after minimum of 2 hours and at latest 24 hours after the first four dosis of ASA
  Groups: Individualized ASA therapy group using platelet inhibition monitoring

SUMMARY:
The aim of this study is to evaluate the incidence of any hemocompatibility related adverse event (HRAE) after LVAD placement in patients responsive to a standard aspirin dose using point-of-care platelet inhibition monitoring compared with initial non-responders who were then up-titrated to achieve a therapeutic response using individualized acetylsalicylic acid (ASA) therapy. Second, to investigate whether patients exhibit temporal changes in ASA sensitivity during LVAD support.

DETAILED DESCRIPTION:
Left Ventricular Assist Device (LVAD) therapy has become a well-established treatment option for end stage heart-failure either as a bridge to transplant or destination therapy. As previously reported, mechanical circulatory support (MCS) has continued to improve patient survival and quality of life due to improvements in device design as well as implantation technique.

However, HRAEs such as stroke, bleeding, and thrombosis, which are consequences of adverse interactions between the pump and circulating blood elements, are associated with the use of LVADs. Despite excellent clinical outcomes of continuous flow LVADs with one-year survival of 83%, the balance of pump thrombosis (PT) and bleeding continues to present a major treatment challenge. Recent reports indicate, that only 80% of the patients supported with the HeartMate 3 (Abbott Inc.) LVAD had a one-year freedom from gastrointestinal bleeding, and freedom from any neurological adverse event. PT is described in up to 8 % of the HeartWare HVAD (Medtronic Inc.) patients and in 1.4% of HeartMate 3 patients.

Therefore, during long-term treatment, oral anticoagulation with vitamin K antagonists (VKA), such as warfarin or phenprocoumon, is essential to reduce HRAEs in LVAD patients. Most recent guidelines of the International Society for Heart and Lung Transplantation (ISHLT) recommend for centrifugal rotary blood pumps (such as the HeartMate 3 and HVAD) to start oral anticoagulation and antiplatelet therapy on post-operative day (POD) 2 or 3, after removal of the chest tubes and an intended target INR of 2.0-3.0. Furthermore, the ISHLT guidelines recommend 81 - 325 mg daily antiplatelet therapy with ASA in addition to warfarin to decrease thrombotic risk. Specifically for HeartMate 3 patients, the manufacturer recommends 81 - 100mg ASA daily therapy which should start 2 or 3 days after implantation. The manufacturer recommended long term oral anticoagulation regimen for the HVAD pump is a combination of warfarin and ASA. In general, ASA should be started at a doses >81mg per day (e.g. moderate-dose ASA of 162mg or high-dose of 325mg per day) within 24 hours after implant if there are no postoperative bleeding complications.

The relevance of these ASA daily dose recommendations for LVAD patients are supported by the results of several recent clinical studies: Najjar et al. identified an ASA daily dose ≤ 81 mg as independent risk factor for HVAD PT; in addition, Teuteberg et al. also identified daily ASA doses ≤ 81 mg as significant risk factor for ischemic and hemorrhagic cerebrovascular accidents. Uriel et al. analyzed HRAEs at 6 months in the Momentum 3 trial (comparing HeartMate II and 3) with antithrombotic management including anticoagulation with warfarin and ASA therapy (81-325 mg daily). Absence of ASA at 30 days was independently associated with development of HRAE or death at 6 months after implantation. Based on these recommendations and recent publications, current best practice at the Medical University of Vienna includes oral anticoagulation with phenprocoumon (INR target of 2.0-2.5) and without contraindication, on POD 3, the antiplatelet therapy with ASA is initiated. ASA daily standard doses vary device-specific from 100 mg (HeartMate 3) to 200 mg (HVAD).

In addition, the optimal antithrombotic regimen remains uncertain, and the frequency of antiplatelet therapy monitoring differs among clinicians.

Several factors contributing to platelet dysfunction may be related to the propensity for bleeding and thrombosis in patients with LVADs. Shear stress may play a role in platelet dysfunction and increase the potential for PT. Acquired von Willebrand factor syndrome may contribute to the bleeding probability in LVAD patients. Other factors that may increase the may increase the risk of LVAD PT include inadequate antithrombotic or anticoagulant therapy, coagulopathy, or platelet disorders. Aspirin resistance is defined as the inability of aspirin to platelet thromboxane A2 production and thus platelet thromboxane A2 and thus reduce platelet activation and aggregation. Thromboxane A2 is synthesized from achidonic acid in several steps. Cyclooxygenase is a key enzyme for this metabolism. ASA inhibits this enzyme, so the platelets are not able to produce Thromboxane A2 anymore. As the platelets have no cell nucleus, they are incapable to resynthesize the Cyclooxygenase so the inhibition lasts their whole life span (approximately seven days).

Numerous studies have shown that aspirin resistance in patients with cardiovascular disease is associated with poor outcomes. Patients with inadequate response to their antiplatelet medications may have a significantly higher risk of myocardial infarction, stent thrombosis, and death. Patients with an excessive response to their antiplatelet agents are at increased risk for bleeding. Recent literature suggests that 30 to 40% of patients on antiplatelet medications may not receive the expected platelet inhibiting effect. Numerous factors may cause inadequate response including: drug interactions (e.g. proton pump inhibitors), genetic differences, pre-existing health conditions (e.g. diabetes) and non-compliance.

Although e.g. the HVAD manufacturer recommends, if ASA alone is the medication chosen for antiplatelet therapy, a check for ASA resistance with a reliable test (e.g., VerifyNow) is recommended to establish the dose or to select an alternative medication, literature comparing outcomes of LVAD patients with standard aspirin therapy (SAT) and dose-adjusted individualized treatment based on platelet inhibition is lacking. Additionally, little is known about etiology, risk factors and outcomes of initial non-responders to ASA therapy after LVAD implantation. To date, there is no standard platelet function test for use in LVAD patients. Karimi et al. adjusted antiplatelet treatment in HeartMate II patients based on thromboelastography, with an aim to achieve normal maximum amplitude. Although light transmission aggregometry (LTA) is considered by many as gold standard for assessing platelet function, ASA responsiveness can be determined by a turbidimetric based optical based assay test (VerifyNow, Accriva Diagnostics).

The main advantage of VerifyNow is its availability as point-of-care testing at any time of the day. No processing of the blood or specialist laboratorian assistant is needed. Several studies covering different topics have shown the benefit of point-of-care testing with the VerifyNow system. Platelet function testing leading to a customized treatment could reduce thrombotic complications in pediatric patients after heart surgery as well as in LVAD-patients or to identify ASA usage before an emergency surgery.

With the VerifyNow ASA responsiveness test, the unprocessed whole blood is automatically transferred in four chambers containing platelet agonists (for example ADP or arachidonic acid) and fibrinogen-coated beads to trigger the activation of the platelets. As the platelets aggregate, the light transmitting through the chambers will increase because the blood sample gets clearer. The device measures the changes in optical signals over a period of a few minutes. The blood of an adequate platelet-inhibited patient forms fewer aggregates allowing less light to pass through in comparison to a blood sample of an inadequate or non-inhibited patient. Results can be expressed in Aspirin reaction units (ARU), which is calculated as a function of the rate and extend of platelet aggregation. Higher ARU reflect a greater arachidonic acid-induced platelet reactivity. The manufacturer defines an ARU ≤ 549 as an evidence of adequate platelet-dysfunction due to aspirin. ARU ≥ 550 indicates no evidence of aspirin-induced platelet dysfunction. Additionally, the platelet activation via P2Y12-receptors can be evaluated with the VerifyNow system. The results are then expressed in P2Y12 Reaction Units (PRU). Values less than 194 PRU are an evidence of a P2Y12-inhibitor effect.

Furthermore, ASA responsiveness not only varies between patients, but it may significantly change within individual LVAD patients also over time. DeNino et al. described two cases, where the patients had been reported to be sensitive to ASA when discharged on POD 10, but during rehospitalization and a repeated test had shown no evidence of aspirin-induced platelet dysfunction. This is in line with a recent study from Morgan et al., were the resistance to ASA increased from 7% at baseline to 32% three months post-implant.

In conclusion, although ASA therapy is routinely recommended in LVAD patients with continuous flow pumps to prevent HRAEs, the substantial number of events despite improved pump designs may call into question the utility of standard ASA doses for all patients and that assessment of individual response to ASA could further improve outcomes and guide therapy in LVAD patients.

ELIGIBILITY:
Inclusion Criteria:

* The participants will be recipients of the routinely used HeartMate 3 (Abbott, Abbott Park, IL) or HVAD (Medtronic Inc., Dublin, Ireland) system implanted at the Medical University of Vienna, which are able and willing to understand and sign the informed consent form, and which do not meet any exclusion criteria.

Exclusion Criteria:

* Age: <18 or >75 years
* Inability to provide informed consent
* No ASA therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of HeartMate 3 LVAD or HVAD recipients implanted at the Medical University of Vienna. Based on the initial ASA response type (responder vs. non-responder) the primary and secondary outcomes will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Freedom from any hemocompatibility related adverse events (HRAEs) in initial ASA responder and initial ASA non-responder. | freedom from any HRAE over 12 months
  The primary question is whether the two groups (initial ASA responder and initial ASA non-responder) differ with regard to freedom from any HRAEs. For this purpose, the Kaplan-Meier curves for the two groups are shown graphically (the graph also shows the number of patients at risk per year). These two curves are compared with each other using a log-rank test. The median freedom from HRAE times are reported separately for both groups, as well as the probabilities according to Kaplan-Meier for different time frames.

SECONDARY OUTCOMES:
Temporal alteration in ASA therapy sensitivity during follow up | change of ASA therapy sensitivity over 3 months
  The null hypothesis of this secondary question is that there is no difference (temporal alteration) in ASA therapy sensitivity during LVAD follow up. We will compare the ARU measured during follow up A and during the next follow up B (3 months later). Depending on distribution of the metric ARU data, the data will be analyzed by a paired t-test or Wilcoxon test. The presence of a normal distribution will be determined with the Shapiro-Wilk-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No